CLINICAL TRIAL: NCT03018249
Title: A Randomized Surgical Window Pilot Investigation of the Relationship of Short Term Medroxyprogesterone Acetate (NSC #26386) Compared to Medroxyprogesterone Acetate Plus Entinostat (NSC #706995) on the Morphologic, Biochemical, and Molecular Changes in Primary Endometrioid Adenocarcinoma of the Uterine Corpus
Brief Title: Medroxyprogesterone Acetate With or Without Entinostat Before Surgery in Treating Patients With Endometrioid Endometrial Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NCI-2017-00058; NCI-2017-00058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY011; NRG-GY011 (Other: NRG Oncology); NRG-GY011 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: FIGO Grade 1 Endometrial Endometrioid Adenocarcinoma; FIGO Grade 2 Endometrial Endometrioid Adenocarcinoma; FIGO Grade 3 Endometrial Endometrioid Adenocarcinoma
MeSH Terms: interventions — entinostat; Hysterectomy; Medroxyprogesterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (medroxyprogesterone acetate, hysterectomy) (Active Comparator): Patients receive medroxyprogesterone acetate IM on day 1 and undergo hysterectomy between days 21-24.
  Interventions: Procedure: Hysterectomy; Other: Laboratory Biomarker Analysis; Drug: Medroxyprogesterone Acetate
- Arm II (medroxyprogesterone acetate, entinostat, hysterectomy) (Experimental): Patients receive medroxyprogesterone acetate IM on day 1 and entinostat PO on days 1, 8, and 15. Patients undergo hysterectomy between days 21-24.
  Interventions: Drug: Entinostat; Procedure: Hysterectomy; Other: Laboratory Biomarker Analysis; Drug: Medroxyprogesterone Acetate

INTERVENTIONS:
Drug: Entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; MS 27-275; MS-275; SNDX-275
  Arms: Arm II (medroxyprogesterone acetate, entinostat, hysterectomy)
Procedure: Hysterectomy — Undergo hysterectomy
  Other Names: Hysterectomy NOS
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Medroxyprogesterone Acetate — Given IM
  Other Names: Amen; Aragest; Ciclotal; Clinofem; Clinovir; Cycrin; Depo-Clinovir; Depo-Provera; Depot-Medroxyprogestereone Acetate; Farlutal; G-Farlutal; Gestapuran; Hysron; Lutoral; Medroxyprogesterone 17-Acetate; Medroxyprogesteroni Acetas; Methylacetoxyprogesterone; Metipregnone; MPA; Nadigest; Nadigest (vet); Nidaxin; Nidaxin (vet); Oragest; Perlutex; Prodasone; Provera; Sodelut G; Veramix

SUMMARY:
This randomized surgical window trial evaluates the effect of adding entinostat to medroxyprogesterone acetate before surgery works on progesterone receptors on endometrioid endometrial tumors. Medroxyprogesterone acetate is a progesterone, a hormone produced by body normally. Entinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving medroxyprogesterone acetate with or without entinostat may effect tumors from endometrioid endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the addition of the histone deacetylase inhibitor, entinostat, in combination with medroxyprogesterone acetate in the pre-operative setting results in up-regulation of activated progesterone receptors (PR) compared to medroxyprogesterone acetate alone.

SECONDARY OBJECTIVES:

I. To assess the response rate (as measured by cellular morphology and proliferation) and change in activated receptor levels with the addition of entinostat at the time of hysterectomy.

OUTLINE: Two arms were randomly allocated to eligible patients with equal probability.

ARM I: Patients receive medroxyprogesterone acetate intramuscularly (IM) on day 1 and undergo hysterectomy between days 21-24.

ARM II: Patients receive medroxyprogesterone acetate IM on day 1 and entinostat orally (PO) on days 1, 8, and 15. Patients undergo hysterectomy between days 21-24.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically proven diagnosis of endometrioid endometrial adenocarcinoma by endometrial curettage or biopsy within 8 weeks prior to registration; central pathology review will be required as part of the study but not for registration purposes
* History/physical examination within 42 +/- 5 days of planned surgical procedure (18-21 days from day 1); further protocol-specific assessments
* The trial is open only to women with primary endometrioid adenocarcinoma of the uterine corpus (all histologic grades and stages) who are planned and appropriate for primary surgical treatment to include removal of the uterine corpus via any surgical modality; the patient must be considered a suitable surgical candidate
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, 2, or 3 within 28 days prior to registration
* Formalin-fixed, paraffin-embedded tumor tissue from the biopsy or curettage must be submitted along with the corresponding pathology report
* Platelets >= 100,000/ul
* Granulocytes (ANC) >= 1,500/ul
* Creatinine =< 1.6 mg/dl
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x upper limits of normal
* Bilirubin within institutional normal limits
* The patient must provide study-specific informed consent and authorization permitting release of personal health information prior to study entry
* Any patients of childbearing potential must have a negative pregnancy test

Exclusion Criteria:

* Patients with any non-endometrioid histology (such as serous, clear cell, or carcinosarcoma)
* Patients who have received prior progestin or anti-estrogen therapy during the 3 months before the diagnosis of endometrioid adenocarcinoma of the uterine corpus is established; estrogen therapy alone is allowed
* Patients with ECOG performance grade of 4
* Patients with history of thrombophlebitis within the past 2 years or ongoing thromboembolic disorders
* Patients who have previously received systemic, radiation or other treatment for uterine cancer
* Patients for whom formalin-fixed, paraffin-embedded tumor tissue from the biopsy or curettage is unavailable
* Patients must not have previously received a non Food and Drug Administration (FDA) approved histone deacetylase (HDAC) inhibitor in a clinical trial setting (entinostat, belinostat)
* Patients must not be currently taking or have ever taken vorinostat (Zolinza, Merck), panobinostat (Farydak, Novartis) or romidepsin (Istodax, Gloucester Pharmaceuticals)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda R Duska, Principal Investigator — NRG Oncology
Locations (234):
- United States (234):
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - John Muir Medical Center-Concord Campus, Concord, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Sacred Heart Hospital, Pensacola, Florida
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Willis-Knighton Medical and Cancer Center, Shreveport, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Spartanburg, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was open to accrual on 8/17/2017. The first patient was enrolled on October 11, 2017. The study closed to accrual 4 months later on 2/9/2018 after 50 patients were enrolled across 13 unique sites.
Groups:
- Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA: Patients receive medroxyprogesterone acetate IM on day 1 and undergo hysterectomy between days 21-24.
- Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat: Medroxyprogesterone acetate IM on day 1 and entinostat PO on days 1, 8, and 15. Followed by hysterectomy between days 21-24.
Period: Overall Study
Arm/Group | Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA | Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA | Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Customized [Count of Participants; unit: Participants]
  30-49 years | 2 | 2 | 4
  50-59 years | 7 | 7 | 14
  60-69 years | 13 | 13 | 26
  70-99 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 24 | 49
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 23 | 22 | 45
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Participants with Endometrioid Cell Type Cancer [Count of Participants; unit: Participants] | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Mean Post-treatment Tumor Progesterone Receptor H-score (Histology Score)
Description: The H-score is defined as the percent cells staining positive (0-100) multiplied by the staining intensity (0, 1, 2 or 3) measured in the tumor by immunohistochemistry and averaged over 3 reviewers. This score can range from 0 to 300. In general, PRs are expected to decrease in response to medroxyprogesterone acetate. It was hypothesized that entinostat would mitigate the decrease in PR relative to the medroxyprogesterone acetate only arm post treatment. Higher PR H-scores post treatment in the arm with entinostat relative to the medroxyprogesterone alone arm would be consistent with this hypothesis. Arm II was thought to result in higher scores which was expected to have a more favorable outcome when treated with MPA therapy.
Time Frame: Specimens were collected at hysterectomy on day 21-24 and analyzed in batch.
Population: Randomized, treated, evaluable specimen. There were 2 participants in each reporting group who withdrew consent prior to treatment; no specimens were submitted for these patients. There were two additional patients with insufficient tumor post-treatment and no slides were submitted; one in each reporting group. There was one additional patient with no specimens submitted in reporting group 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA | Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat
Number analyzed (Participants) | 22 | 21
units on a scale | 53.6 (64.8) | 42.7 (49.0)
Statistical Analysis 1: Comparison: Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA vs Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat; Test type: Superiority; p = 0.87, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percentage of Participants With a Histologic Response
Description: Pre- and post-treatment slides for each patient were evaluated in pairs for complete or partial histologic response by one reviewer. Pre- and post-treatment slides for each patient were evaluated in pairs for complete or partial histologic response by one reviewer. A histologic response was defined as either the absence of identifiable adenocarcinoma in the hysterectomy specimen section (complete) or, subjectively, as the presence of a complex proliferation of glands that retain the architectural characteristics of adenocarcinoma, but with features of secretion, decreased nuclear stratification, or the presence of eosinophilic, squamous or mucinous metaplasia, when this was absent in the initial sample (partial).
Time Frame: Specimens were collected at initial diagnostic biopsy and at hysterectomy on day 21-24 and analyzed in batch.
Population: Randomized, treated, evaluable pre and post treatment specimen available. There were 2 participants in each reporting group who withdrew consent prior to treatment; no specimens were submitted for these patients. There was one participant with an inevaluable pre-treatment slide. There were two additional patients with insufficient tumor post-treatment and no slides were submitted; one in each reporting group. There was one additional patient with no specimens submitted in reporting group 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA | Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat
Number analyzed (Participants) | 22 | 20
Participants | 16 | 14
Statistical Analysis 1: Comparison: Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA vs Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat; Test type: Superiority; Mean Difference (Final Values) = 2.7, 95% CI 2-sided [-25 to 30]

3. Secondary Outcome: Percent of Participants With a Ki67 Response
Description: A response was defined as a decrease in Ki-67 protein expression in tumor from pre- to post-treatment.
Time Frame: Specimens were collected at initial diagnostic biopsy and at hysterectomy on day 21-24 and analyzed in batch.
Population: Randomized, treated, evaluable pre and post treatment specimens available. There were 2 participants in each reporting group who withdrew consent prior to treatment; no specimens were submitted for these patients. There was one participant with an inevaluable pre-treatment slide. There were two additional patients with insufficient tumor post-treatment and no slides were submitted; one in each reporting group. There was one additional patient with no specimens submitted in reporting group
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA | Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat
Number analyzed (Participants) | 22 | 20
Participants | 15 | 18
Statistical Analysis 1: Comparison: Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA vs Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat; Test type: Superiority; Mean Difference (Final Values) = 21.8, 95% CI 2-sided [-16.7 to 45.3]

4. Secondary Outcome: The Frequency and Severity of CTCAE Version 4.0 Graded Adverse Events (AE)
Description: Maximum grade of physician assessed adverse events reported during treatment and up to 45 days after surgery. Grades start with 1 which is considered mild through grade 5 which is death. Participants on this study had adverse event grades up to grade 3 which is considered moderately severe.
Time Frame: Up to 45 days after surgery
Population: Eligible and Treated Patients
Measure: Number; unit: participants
Arm/Group | Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA | Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat
Number analyzed (Participants) | 23 | 23
participants
  Grade 1 AE | 11 | 9
  Grade 2 AE | 4 | 6
  Grade 3 AE | 2 | 2
  Grade 4 AE | 0 | 0
  Grade 5 AE | 0 | 0

5. Other Pre Specified Outcome: Mean Post-treatment Tumor Estrogen Receptor Score
Time Frame: Up to 3 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Co-expression of PR, Ki67, and p21
Description: Will be compared between the arms.
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From initiation of treatment up to 45 days post-surgery
Description: There were 2 participants in each reporting group who withdrew consent prior to treatment; no specimens were submitted for these patients. No AEs were reported.
Arm/Group | Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA | Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/23 | 1/23
Other Adverse Events (participants affected / at risk) | 14/23 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA (N=23) | Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat (N=23)
Thromboembolic Event (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Skin infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Medroxyprogesterone Acetate, Hysterectomy) MPA (N=23) | Arm II (Medroxyprogesterone Acetate, Entinostat, Hysterectomy) MPA and Entinostat (N=23)
Anemia (Blood and lymphatic system disorders) | 3 | 3
Abdominal Pain (Gastrointestinal disorders) | 4 | 8
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhea (Gastrointestinal disorders) | 2 | 4
Dry Mouth (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 4
Edema Limbs (General disorders) | 3 | 2
Fatigue (General disorders) | 4 | 8
Injection Site Reaction (General disorders) | 4 | 5
Pain (General disorders) | 4 | 4
Neutrophil Count Decreased (Investigations) | 0 | 2
Platelet Count Decreased (Investigations) | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 3 | 1
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 2
Urinary Incontinence (Renal and urinary disorders) | 2 | 0
Pelvic Pain (Reproductive system and breast disorders) | 2 | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 4
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Hypertension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT03018249/Prot_SAP_000.pdf